CLINICAL TRIAL: NCT06381869
Title: Study of Comparative Bioavailability, Randomized, in Open Cross Over the Kinetics of Subsequent Plasma Amino Acid Concentrations the Consumption of Pea Protein "NUTRALYS ® S85 Plus".
Brief Title: Bioavailability of Pea Protein in Young and Old Volunteers
Acronym: NUTRALYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roquette Freres (Industry)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government); Université d'Auvergne (Other)
Responsible Party: Principal Investigator, Ruddy Richard, Director of the Nutrition Exploration Unit, Clinical professor, Université d'Auvergne
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CRNHA 2018-2
Record Dates: First submitted 2024-04-16; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Healthy Male Volunteers
Keywords: Protein; Bioavailability; Pea protein; Amino acidemia
MeSH Terms: interventions — Pea Proteins; Whey Proteins; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young volunteers (Other): Volunteers under 30 years old
  Interventions: Dietary Supplement: Pea protein (NUTRALYS ® S85 plus) in water; Dietary Supplement: Pea protein (NUTRALYS ® S85 plus) within meal; Dietary Supplement: Whey protein in water; Dietary Supplement: Whey protein within meal
- Elderly volunteers (Other): Volunteers over 65 years old.
  Interventions: Dietary Supplement: Pea protein (NUTRALYS ® S85 plus) in water; Dietary Supplement: Pea protein (NUTRALYS ® S85 plus) within meal; Dietary Supplement: Whey protein in water; Dietary Supplement: Whey protein within meal

INTERVENTIONS:
Dietary Supplement: Pea protein (NUTRALYS ® S85 plus) in water — After selection and randomization, the subjects will consume per os Pea protein (NUTRALYS® S85 plus) in water containing 0,41 g of tested protein/kg of body weight.
Dietary Supplement: Pea protein (NUTRALYS ® S85 plus) within meal — After selection and randomization, the subjects will consume per os Pea protein (NUTRALYS® S85 plus) within a meal containing 0,41 g of tested protein/kg of body weight.
Dietary Supplement: Whey protein in water — After selection and randomization, the subjects will consume per os whey protein in water containing 0,41 g of tested protein/kg of body weight.
Dietary Supplement: Whey protein within meal — After selection and randomization, the subjects will consume per os whey protein within a meal containing 0,41 g of tested protein/kg of body weight.

SUMMARY:
The aim of this study done in healthy, non-malnourished young and elderly subjects, is to measure the bioavailability of protein intake and the variation of metabolic markers following consumption of pea protein " NUTRALYS ® S85 plus" or a reference protein brought in water either alone or at the end of a standardized meal.

ELIGIBILITY:
Inclusion Criteria:

* Adult male volunteers, aged over 65 or under 30
* Body mass index (weight in kg/ height² in m²) between 22 and 28 kg/m²,
* Subjects considered to be healthy by the principal investigator doctor according to the interview, medical and clinical examination,
* Biological assessment considered compatible with participation in the study,
* Persons able to sign the informed consent,
* Persons affiliated to social security scheme.

Exclusion Criteria:

* Pathologies or treatments not compatible with the study
* Food allergy or a contraindication to the consumption of the products tested
* Subject in a situation which, in the opinion of the investigator, could interfere with their optimal participation in the study or constitute a particular risk for the subject,
* Subject with a particular diet (vegetarians, vegans, nutritional supplements, etc.),
* Subject weighing < 55 kg,

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
Leucine blood concentration | 0 minute before eating the test meals, then regularly until 360 minutes after ingestion.

SECONDARY OUTCOMES:
Essential amino acids blood concentration (µmol/L) | 0 minute before eating the test meals, then regularly until 360 minutes after ingestion.
Non essential amino acid blood concentration (µmol/L) | 0 minute before eating the test meals, then regularly until 360 minutes after ingestion.
Blood glucose concentration (g/L) | 0 minute before eating the test meals, then regularly until 360 minutes after ingestion.
Blood insulin concentration (μIU/ml) | 0 minute before eating the test meals, then regularly until 360 minutes after ingestion.
Blood lipid profile (glycerol concentration in mg/l and non-esterified fatty acids concentration in mg/l) | 0 minute before eating the test meals, then regularly until 360 minutes after ingestion.
Blood inflammatory profile (TNF-α blood concentration in pg/ml and IL-6 blood concentration in pg/ml) | 0 minute before eating the test meals, then regularly until 360 minutes after ingestion.

CONTACTS AND LOCATIONS:
Locations (1):
- Unité d'Exploration en Nutrition Centre de Recherche en Nutrition Humaine d'Auvergne, Clermont-Ferrand, France